CLINICAL TRIAL: NCT03601767
Title: Derivation and Validation of a Prognostic Model for Septic Patients at Hospital Admission
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera San Paolo (Other)
Responsible Party: Principal Investigator, Livio Colombo, Consultant in Acute Medicine, Azienda Ospedaliera San Paolo
Other Study IDs: 38788/2017
Record Dates: First submitted 2018-05-30; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Sepsis
Keywords: sepsis; score
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the present study is to develop a prognostic tool to assess the risk of dead and major complications in patient admitted to hospital for infection. A detailed database of clinical, biochemical and microbiological data is recorded and each item is analyzed and compared with clinical outcomes to develop a prognostic score.

ELIGIBILITY:
Inclusion Criteria:

* al least 18 years old
* admission to hospital for any infection for more than 72 hours

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects presenting to the accident and emergency department and admitted to hospital for any infection
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-09-20 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
mortality | at 28 days

SECONDARY OUTCOMES:
major complications | at 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Paolo Polo Univesitario - ASST Santi Paolo e Carlo, Milan, Italy